CLINICAL TRIAL: NCT02590419
Title: Application of Diffusion Tensor Imaging and Tractography in Epilepsy Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Andrew Parrent (Other)
Collaborators: University of Western Ontario, Canada (Other); Synaptive Medical (Industry)
Responsible Party: Sponsor-Investigator, Andrew Parrent, Neurosurgeon; Associate Professor, London Health Sciences Centre
Organization: London Health Sciences Centre (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UWO HSREB Ref#10317
Record Dates: First submitted 2015-07-08; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Temporal Lobe Epilepsy
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Control Group (involvement of BrightMatter™ Plan (BMP)): Patients with temporal lobe epilepsy, who have been identified as candidates for anterior temporal lobe resection (ATLR) will be recruited. All epilepsy patients will have clinical MRI scans that include a diffusion tensor imaging (DTI) protocol. Surgery will be carried out according to usual standard of care, without the use of processing for DTI tractography. Additional clinical scanning with the same protocol will be carried out post-operatively at 6 months. Pre-operative and post-operative (6-month) visual field assessments (Estermann Perimetry and Humphrey Perimetry) will also be carried out . Primary outcomes will be assessed to identify the baseline incidence of visual of postoperative visual field deficits.
- Treatment Arm (Experimental): Treatment group (involvement of all three products BrightMatter™ Plan (BMP), BrightMatter™ Bridge (BMB), and BrightMatter™ Guide(BMG): A treatment group (prospective enrollment) that uses the interventional technology will be recruited based on the same eligibility criteria as control cohort. All epilepsy patients will have clinical MRI scans that include a DTI protocol. For this treatment group of patients, the BrightMatter system (BMB,BMP, and BMG) will be employed pre-operatively and intra-operatively for planning before and guidance during anterior temporal lobe resection (ATLR). Additional clinical scanning with the same protocol will be carried out post-operatively at 6 months. Pre-operative and post-operative (6-month) visual field assessments (Estermann Perimetry and Humphrey Perimetry) will also be carried out. Primary outcomes will be assessed to evaluate the effect of surgical planning and guidance with DTI tractography on outcomes, by comparison against the control cohort.
  Interventions: Device: BrightMatter™ products

INTERVENTIONS:
Device: BrightMatter™ products — BrightMatter™ Plan (BMP): BMP is a software that enables surgeons to plan their neurosurgery preoperatively. BMP automatically generates whole brain tractography and highly accurate fusion of anatomical MRI and DTI images.
  BrightMatter™ Bridge (BMB):BMB involves offering SMI's MRI expertise to ensure a smooth workflow in neuroimaging including DTI to ensure optimized protocols are used to acquire the DTI images. Once the images are acquired, they are evaluated for their quality in real time using a quality control (QC) algorithm. The QC allows quality assessment of DTI images at the time-of-scan allowing for immediate correction while the patient is still there and reduces the need for patient re-scan.
  BrightMatter™ Guide (BMG): BMG is a neuro-navigation system that utilizes the DTI information and the trajectory planned by the surgeon in BMP pre-operatively, but bringing it into the operating room intraoperatively.
  Other Names: BrightMatter™ Plan, BrightMatter™ Bridge, BrightMatter™ Guide
  Arms: Treatment Arm

SUMMARY:
Using Synaptive Medical's BrightMatter™ products to better visualize and plan epilepsy surgeries by considering white matter tracts, and considering whether the technology results in improved clinical outcomes.

DETAILED DESCRIPTION:
A common goal of focal brain resection is the removal of a lesion while preserving healthy eloquent tissues of the brain. One such eloquent area that is commonly aimed to be preserved are the white matter nerve fiber tracts which is critical of brain communication and function. This study aims to investigate whether the use of Synaptive Medical's BrightMatterTM technology can help neurosurgeons to better visualize and plan surgeries by considering the white matter tracts, and whether it results in improved clinical outcomes. This study will investigate the preservation of the optic radiations in anterior temporal lobectomy epilepsy surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with temporal lobe epilepsy between 18 and 65 years of age.
* Patients whose seizures are disabling and/or are not controlled by any form of epileptic medication.
* Patients whose clinical pre-surgical investigations indicates the need for anterior temporal lobe resection (ATLR).

Exclusion Criteria:

* Prior resective epilepsy surgery.
* Past or planned non resective epilepsy surgery (such as a corpus callosotomy and vagal nerve stimulator placement).
* Contraindication to MRI, and/or whom are (or suspect to) being pregnant.
* Complicated medical problems such as cancer or heart disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Total volume of tract damage | Assessed between pre and post-operative visits (6 month follow-up).
  Tract damage
Resection Zone | Assessed at surgical visit
  Identification of resected region
Post-operative visual field testing | Assessed at post-operative visit (6 month follow-up)
  Outcome will be measured using a routine visual field testing procedure known as the Humphrey and Estermann perimetry test.

SECONDARY OUTCOMES:
Total neurological planning time | Assessed during planning phase of surgery, between both pre and post-operative visits (6 month follow-up).
  Measured in hours
Total OR time | Assessed during surgical visit
  Measured in hours
Duration of hospital stay | Assessed during surgical visit up to 26 weeks.
  Measured in # of days
Number of seizure free days | Assessed between surgical date until post-operative visit (6 month follow-up).
  Measured in # of days
Total cost of surgery | Assessed through study completion, an average of 1 year.
Quality of life assessment | Assessed during surgical visit up to 26 weeks.
  Measured using a standard epilepsy questionnaire known as the WHOQOL-BREF questionnaire (World Health Organization Quality of Life Assessment (WHOQOL-BREF))
Functional impairment | Assessed during surgical visit up to 26 weeks.
  Measured using a routine functional impairment test known as the Karnofsky performance scale
Morbidity and complications | Assessed through study completion, an average of 1 year.
  Number of cases
Seizure control after surgery | Assessed at surgical visit up to 26 weeks.
  Assessed using a routine seizure control test known as the Engel score, assessed by a neurologist/epileptologist

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Parrent, Principal Investigator — London Health Sciences